CLINICAL TRIAL: NCT06393933
Title: Oral Health Knowledge, Attitude and Behaviour Among Preclinical and Clinical Dental Students: A Cross Sectional Study On A Sample of Adult Egyption Students.
Brief Title: Oral Health Knowledge, Attitude and Behaviour Among Preclinical and Clinical Dental Students
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Emad Ahmed, Principle investigator, Cairo University
Other Study IDs: 20122
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Oral Health Knowledge

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Oral health knowledge is considered to be an essential prerequisite for oral health related attitude and behavior. Attitude is a mirror of individuals' beliefs, experiences, perception of the cultures, and social interactions. Basically, positive health attitude means positive health behavior. This also applies to a great extent to oral health attitude and is of paramount importance when it relates to oral health professionals. Therefore, with proper knowledge and oral health behaviour, oral health professionals can play an important role in oral health education of their patients as well as act as role models for these patients and community at large.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), oral health problems are still not well controlled globally despite the considerable improvements in oral health measures among populations. This state of oral health might be related to the rapid development of oral diseases following lifestyle changes such as consumption of a sugar-rich diet, lack of water fluoridation, and other socio-environmental factors. The high incidence and prevalence of oral diseases globally qualifies oral health as a serious public health issue. In addition, oral disease treatments are considered to be the fourth most expensive disease treatments in most industrial countries. That makes oral health a huge burden at both the individual and the community level. Oral disease is a worldwide epidemic and has imposed an enormous burden on the health and economy of the whole society. The number of people with untreated oral conditions worldwide increased from 2.5 million in 1990 to 3.5 billion in 2015, with a 64.0% increase in disability-adjusted life years due to oral conditions. Among these conditions, untreated dental caries, severe periodontitis, and missing teeth are the three most common and chronic 3 infectious oral diseases. Fortunately, most oral diseases, especially dental caries and periodontal diseases, are largely preventable through various promotion interventions. Oral health education (OHE) was once considered the most cost-effective intervention.

Oral health is considered an important component of general health that has been shown to influence the quality of life. Oral health may affect the individual's appearance, social functions, and physical and psychological daily activities. Periodontal health is a major component of oral health that concentrates on the prevention of inflammatory diseases in supportive tissue surrounding the teeth. Oral hygiene practice can be defined as any effort performed by the individual to remove supra-gingival biofilm. Studies have shown that poor oral hygiene will lead to gingival inflammation and have established a linear relationship between plaque development and the presence of gingivitis. The development of gingivitis had been linked to the development of periodontitis. Therefore, cleaning the oral cavity is essential because it removes bacterial accumulation and prevents periodontal disease progression. Dental students are the future leaders in oral health care and are expected to be teachers of oral hygiene as well as role models of self-care regimens for their patients as their dental education progresses. In a dental school setting, it is critical to evaluate yearly progress of dental students learning about self-care regimens such as oral health attitudes and behavior.

The Egyptian dental education model defines a strong preclinical-clinical contrast.

Furthermore, it implements discipline-based curricula, in which large-group educational lectures and apprenticeship methods of clinical training are the primary methods of teaching. This sharp transition from the preclinical to the clinical phases of education has profound effects on dental students, as they shift from their function as recipients of theoretical oral hygiene education to becoming contributors and educators themselves in charge of actual patients' oral health.

The Hiroshima University-Dental Behavioural Inventory (HU-DBI), developed by Kawamura, has been frequently used to assess university students' oral health-related knowledge, attitudes, and behaviours due to its high psychometric properties that associate students' replies with clinical outcomes, including dental caries and periodontal diseases. It consists of twenty questions eliciting dichotomous responses (agree/disagree).

During the last 30 years, the HU-DBI has been used by dental researchers in more than 10 European countries, including Belgium, Croatia, Finland, France, Germany, Greece, Italy, Lithuania, Turkey, and the United Kingdom. In addition, the HU-DBI has been translated from Japanese into English, Finnish, Chinese, Korean and Arabic for cross-cultural comparisons. The study aims at evaluating the Oral Health Knowledge, Attitude and Behaviour of Preclinical and Clinical Adult Egyptian Dental Students enrolled at the faculty of dentistry, Cairo University using a modified Hiroshima University-Dental Behaviour Inventory (HUDBI) survey.

ELIGIBILITY:
Inclusion Criteria:

1. Preclinical dental students included from 1st and 2nd academic years.
2. Clinical dental students included from 4th and 5th academic years.
3. Medically free dental students.

5- Provide informed consent

Exclusion Criteria:

1. Dental students at 3rd dental year that are not fulfilling the full criteria to be examined.
2. The postgraduate students and residents.
3. Students that are having problem in opening their mouth or undergoing intermaxillary fixation where oral examination will not be possible

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Preclinical and clinical dental students will be recruited in a consecutive manner from a clinic of periodontology, Faculty of Dentistry, Cairo University, following a predetermined appointments.A full survey will be filled for each student. Before filling the survey, the aim of the study will be explained to each student and the student's acceptance to participate in the survey will be receiveThe survey will be filled through a face-to-face personal interview with the student using simple questions.Clinical oral health examination will be held on a dental unit using the light of the unit, mirror and WHO periodontal probe. Also the socioeconomic status scale will be filled; the scale of Fahmy and El-Sherbini was originally published 1983.
Sampling Method: Probability Sample
Enrollment: 546 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
oral health knowledge | 3 months
  It will be assessed by Modified Hiroshima University-Dental Behavioural Inventory (HU-DBI) survey and dependent on items no. 2, 8, 10, 15, and 19.

SECONDARY OUTCOMES:
Oral health attitude and behaviour | 3 months
  that will be assessed by Modified Hiroshima University- Dental Behavioural Inventory (HU-DBI) survey. Oral health attitudes score was dependent on items no. 6, 11, and 14, and behaviours score on items no. 4, 9, 12, and 16.
- Socioeconomic Status | 3 months
  It assessed by Updated Socioeconomic Status Scale for Health Research.
Clinical oral health assessment | 3 months
  s component and calculus component